CLINICAL TRIAL: NCT06850818
Title: Endoprosthesis Registry Heidelberg (EPR-HD): Registry for the Analysis of Patients Following Primary Implantation or Revision Surgery of Artificial Joints in Hip and Knee Joint Pathologies
Brief Title: Heidelberg Registry for Hip and Knee Joint Implants and Revisions
Acronym: EPR-HD
Status: Recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Mustafa Hariri, Principal Investigator, University Hospital Heidelberg
Other Study IDs: S-003/2025
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis; Arthroplasty
Keywords: Endoprostheses; Arthroplasty; Joint Replacement; Osteoarthritis; Registry; Knee; Hip
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Endoprosthesis Registry Heidelberg (EPR-HD) is a clinical registry designed to systematically collect and analyze data from patients undergoing primary implantation or revision surgery of artificial hip and knee joints. The main objective of the registry is to evaluate long-term outcomes, complication rates, implant survival, and functional results associated with joint replacement procedures in patients with various hip and knee joint pathologies.

By gathering comprehensive clinical data, EPR-HD aims to improve the understanding of patient outcomes after endoprosthetic procedures, identify potential factors influencing implant success, and support evidence-based improvements in surgical techniques and patient care. The registry includes adult patients treated at Heidelberg University Hospital, with data collected at multiple time points during routine clinical follow-up. This registry will contribute to the optimization of joint replacement strategies and promote high-quality patient care.

DETAILED DESCRIPTION:
The Endoprosthesis Registry Heidelberg (EPR-HD) is designed to provide comprehensive, long-term data on patients undergoing primary implantation or revision surgery of hip and knee endoprostheses. The registry aims to enhance the understanding of factors affecting the survival and functionality of joint implants, providing essential insights for optimizing surgical strategies and improving patient outcomes.

Hip and knee arthroplasty are among the most common orthopedic procedures worldwide, yet long-term data on implant performance and patient-specific risk factors remain limited. The EPR-HD registry addresses this knowledge gap by systematically collecting clinical data, including patient demographics, surgical details, implant characteristics, perioperative outcomes, and long-term follow-up results. Complication rates, reasons for revision, and functional outcomes such as mobility, pain levels, and quality of life will be assessed over time.

The registry includes adult patients treated at Heidelberg University Hospital who undergo either primary implantation or revision surgery of hip or knee joints due to various pathologies, including osteoarthritis, rheumatoid arthritis, and post-traumatic conditions. Data will be collected prospectively during routine clinical visits at standardized follow-up intervals (e.g., 1 year, 3 years and every 5 years postoperatively).

By evaluating real-world clinical outcomes, EPR-HD will contribute to identifying risk factors associated with implant failure and complications, supporting the development of evidence-based treatment protocols. The insights gained from this registry will promote high-quality care, optimize surgical decision-making, and improve the long-term success of joint replacement procedures in diverse patient populations

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing hip or knee arthroplasty at our institution
* All patients undergoing revision surgery following hip oder knee arthroplasty

Exclusion Criteria:

* Lack of prospective consent for study participation
* Lack of capacity to provide informed consent
* Minor status (underage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery at the Department of Orthopedic Surgery, Heidelberg University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Survival analysis with the endpoint revision for any reason | Preoperative, 1 year, 3 years, and every 5 years
  Kaplan Meier Analysis

SECONDARY OUTCOMES:
Knee Society Score | preoperative, 1 year, 3 years and every 5 years
  The Knee Society Score (KSS) provides a 0 to 100 score measuring function, pain, and range of motion in the knee before and after surgery. A score of 0 indicates the worst outcome, while a score of 100 indicates the best outcome.
Forgotten Joint Score | preoperative, 1 year, 3 years and every 5 years
  The Forgotten Joint Score assesses how aware the patient is of their joint in everyday life. A score of 0 is the worst (always aware) while a score of 100 is the best (the patient is so comfortable, they forget that the joint was replaced).
Oxford Knee/Hip Score | preoperative, 1 year, 3 years and every 5 years
  The Oxford Knee Score (OKS) provides a 0 to 48 score measuring function, pain, and range of motion in the knee before and after surgery. A score of 0 indicates the worst outcome, while a score of 48 indicates the best outcome
Harris Hip | preoperative, 1 year, 3 years and every 5 years
  This survey assesses pain, deformity, and range of motion of the hip. A score of 0 indicates the worst outcome and 100 indicates the best.
Tegner Activity Scale | preoperative, 1 year, 3 years and every 5 years
  The Tegner Activity Scale is a standardized scoring system used to assess a patient's level of physical activity and participation in sports or occupational tasks. The scale ranges from 0 to 10, where 0 indicates disability due to knee problems and 10 represents participation in competitive sports at the national or international elite level
The University of California, Los Angeles (UCLA) Activity Score | preoperative, 1 year, 3 years and every 5 years
  The University of California, Los Angeles (UCLA) Activity Score is a validated scale used to assess the activity level of patients, particularly following joint replacement surgeries. The score ranges from 1 to 10, where 1 represents complete inactivity and dependence on others, while 10 indicates regular participation in impact sports.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No